CLINICAL TRIAL: NCT00068211
Title: A Phase II Study of ILX651 Administered Intravenously Daily for Five Consecutive Days Once Every 3 Weeks in Patients With Inoperable Locally Advanced or Metastatic Melanoma.
Brief Title: Study of ILX651 in Patients With Inoperable Locally Advanced or Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILX651-211
Record Dates: First submitted 2003-09-09; First posted 2003-09-11 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Melanoma
Keywords: Metastatic Melanoma; Melanoma; Inoperable Locally Advanced Melanoma
MeSH Terms: conditions — Melanoma | interventions — tasidotin

INTERVENTIONS:
Drug: ILX651

SUMMARY:
This is a Phase II, non-randomized, open label study of ILX651 in patients with inoperable locally advanced or metastatic melanoma. Approximately 60 patients will be enrolled in this study that is expected to last 18 months. All patients will be treated with ILX651 administered IV daily for 5 consecutive days once every 21 days. The primary objective of this study is to determine the overall response rate for all patients who are treated with ILX651. The secondary objectives are to determine the progression free survival at 18 weeks, duration of response, time to tumor progression, survival, safety/tolerability of ILX651 and to evaluate the pharmacokinetic profile.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed inoperable locally advanced or metastatic malignant melanoma.
* Measurable disease. Measurable lesions should be outside the field of radiation. Where measurable lesions are within a previously irradiated field, there must be objective evidence of progression of the lesion prior to patient enrollment.
* Male or female patients greater than or equal to 18 years of age.
* ECOG performance status of 0 or 1.
* Must have adequate organ and immune system function as indicated by the following laboratory values, obtained less than or equal to 2 weeks prior to registration: A. Absolute neutrophil count(ANC) greater than or equal to 1.5 x 1,000,000,000. B.Hemoglobin greater than or equal to 9.0 g/Dl. C. Platelet count greater than or equal to 100 x 1,000,000,000/L. E. Serum creatinine or calculated creatinine clearance less than or equal to 1.5 mg/dL or greater than or equal to 60 mL/min. F. Serum total bilirubin less than or equal to 2.0 mg/dL. G. AST and ALT less than or equal to 3 times the upper limit of normal (ULN) OR less than 5 times the ULN if secondary to liver metastases. H. Alkaline phosphatase less than or equal to 5 times the ULN (unless bone metastases are present in the absence of liver metastases).
* Anti-cancer therapy, major surgery, or irradiation must have been completed at least 4 weeks before enrollment in this study. Patient must have recovered from the acute side effects incurred as a result of previous therapy.
* Female patients with childbearing potential must have a negative pregnancy test within 7 days of study enrollment. Men and women of reproductive potential must use an effective contraceptive method while enrolled in the study.
* Signed informed consent (includes HIPAA authorization).

Exclusion Criteria:

* Patients with uncontrolled congestive heart failure or angina, patients with a history of myocardial infarction within 2 months of enrollment, or patients with cardiac functional capacity Class III or IV as defined by the New York Heart Association Classification.
* Previously treated with systemic chemotherapy.
* Prior radiotherapy to the only site of measurable disease.
* Known hypersensitivity to study drug or its analogs.
* Active ocular melanoma. Patients with a primary diagnosis of ocular melanoma will not be excluded provided the primary ocular melanoma is no longer present and the recurrence is distal.
* Use of investigational agents within previous 30 days.
* Known, active infection, or known HIV positive or presence of an AIDS related illness.
* Active secondary malignancy.
* Presence of symptomatic active brain metastases, including leptomeningeal involvement. Prior evidence of brain metastasis is permitted only if the patient has been in clinical complete remission for at least 1 month after therapy.
* Uncontrolled hypertension. Patients with hypertension must have their blood pressure controlled on antihypertensive medications as assessed by the investigator.
* Patients with prior radiation therapy to greater than 25% of the bone marrow (eg, no whole pelvic irradiation is allowed).
* Any significant concurrent disease or illness, or psychiatric disorders or alcohol or chemical abuse that would, in the opinion of the investigator, compromise patient safety or compliance, or interfere with the interpretation of study results.
* Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-08; Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Arizona Cancer Center at Scottsdale, Scottsdale, Arizona
  - Univ of Arizona Cancer Center, Tucson, Arizona
  - USC / Norris Cancer Center, Los Angeles, California
  - Cancer Institute Medical Group, Santa Monica, California
  - Univ of Colorado Cancer Center/ Anschutz Cancer, Aurora, Colorado
  - US Oncology / Cancer Centers of Florida, Orlando, Florida
  - US Oncology / Kansas City Oncology, Overland Park, Kansas
  - Beth Israel Medical Center, Boston, Massachusetts
  - US Oncology / Kansas City Oncology and Hematology, Kansas City, Missouri
  - Center for Cancer Care Research, St Louis, Missouri
  - US Oncology / Albany Regional Cancer Center, Albany, New York
  - US Oncology / Dayton Oncology and Hematology, Kettering, Ohio
  - US Oncology / Cancer Centers of the Carolinas, Greenville, South Carolina
  - US Oncology / Mary Crowley Medical Research, Dallas, Texas
  - US Oncology /Texas Oncology, Fort Worth, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - US Oncology/ Tyler Cancer Center, Tyler, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - US Oncology / Cancer Care Northwest, Spokane, Washington